CLINICAL TRIAL: NCT03025334
Title: Transcranial Direct Current Stimulation Treatment of Cognitive Dysfunction in Parkinson's Disease
Brief Title: tDCS on Parkinson's Disease Cognition
Acronym: tDCS-PD-fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Parkinson Society Canada (Other)
Responsible Party: Principal Investigator, Ji Hyun Ko, PhD, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2016:052
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham tDCS (Sham Comparator): sham tDCS (30sec ramp-up and 3sec ramp-down)
  Interventions: Device: High-definition transcranial direct current stimulation
- Real tDCS right (Active Comparator): Real anodal tDCS (right DLPFC)
  Interventions: Device: High-definition transcranial direct current stimulation

INTERVENTIONS:
Device: High-definition transcranial direct current stimulation — brain stimulation to increase neuronal excitability in the targeted regions

SUMMARY:
Parkinson's disease (PD) has been classically regarded as a "movement disorder", so earlier work has focused on treating motor symptoms only. As PD patients now have longer life expectancy, the relatively slowly progressing cognitive deficits (compared to their motor deficits) have become one of the major challenges. Approximately 80% of PD patients eventually become demented. Therefore cognitive dysfunction is one of the most significant factors affecting the quality of life of patients with PD. While dementia in Parkinson's disease is routinely treated by cholinesterase inhibitors (e.g., donepezil and rivastigmine), their efficacy on mild cognitive impairment found in non-demented PD is questionable. Alternative approaches have been proposed including transcranial direct current stimulation (tDCS) but no consensus has been reached. This can be attributed mainly to: (1) imprecise knowledge of the underlying functional circuitry mediating this disease manifestation and (2) inter-individual variability. Here, the investigators will utilize a novel personalized network analysis approach to elucidate on the underlying mechanisms of the effect of tDCS on cognitive dysfunction in non-demented PD patients.

It has been well documented that the caudate nucleus plays an important role in cognitive dysfunction found in PD. In the investigators' preliminary resting-state functional magnetic resonance imaging (fMRI) study, they have shown that the connectivity of the right caudate nucleus is correlated to cognitive status of PD patients measured by the Montreal Cognitive Assessment (MoCA). The investigators hypothesize that tDCS on the left and/or right dorsolateral prefrontal cortex may restore the functional connectivity of the right caudate nucleus which may in turn improve patients' cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet diagnostic criteria for idiopathic Parkinson's disease, defined as the presence of two or more of the cardinal clinical features of PD in the absence of known causes of parkinsonism such as encephalitis or neuroleptic treatment
* Ability to provide written informed consent
* defined by the Diagnostic and Statistical Manual of Mental Disorders; DSM-5)
* Age > 40
* fluent in English.
* Patients' cognitive statuses will be evaluated by the participating neuropsychiatrist or a trained psychiatry or neurology resident.

Exclusion Criteria:

* Patients with dementia (defined as a Montreal Cognitive Assessment score < 18)
* Atypical parkinsonian features including myoclonus, apraxia, oculomotor abnormalities, ataxia, sensory loss, or pyramidal signs.
* Abnormal MRI
* metal implants or a cardiac pacemaker
* Pregnant or breastfeeding women (female subjects of child bearing potential will be screened for pregnancy before MRI imaging).
* severe dyskinesia that may interfere with the quality of the scan (e.g., dyskinesia involving head movement).
* severe hypertension.
* cardiovascular disease.
* Patients with a history of seizure, stroke, moderate to severe head injury, high intracranial pressure, severe headaches, or presence of other neurologic disease that may be associated with an altered seizure threshold; or concurrent medication use, such as tricyclic antidepressants, neuroleptic medications, or other drugs that are known to lower seizure threshold
* secondary conditions that may significantly alter electrolyte balance or lower seizure threshold.
* Family history of epilepsy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
cognitive performance in neuropsychological tests | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada